CLINICAL TRIAL: NCT04512599
Title: Short Chain Fatty Acid Enhancing Prebiotics and Normalization of Parkinson's Disease Microbiome: A Pilot Tolerability Study
Brief Title: Prebiotics in the Parkinson's Disease Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Deborah Hall, MD, Professor of Neurological Sciences, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ORA20072703
Record Dates: First submitted 2020-07-31; First posted 2020-08-13 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
Keywords: microbiome; prebiotic
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study is an open-label, non-randomized study in Parkinson's disease participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Open-label consumption of prebiotic bar(s); 1 bar for 3 days; followed by 2 bars for 7 days
  Interventions: Other: Prebiotic Bar

INTERVENTIONS:
Other: Prebiotic Bar — The prebiotic bar is a proprietary formula created by the study co-investigators, who will not be involved in participant recruitment, selection or outcome measures.The prebiotic bars will be shipped and stored at room temperature prior to consumption.

SUMMARY:
There are about one million Parkinson's disease (PD) patients in America. The risks associated with whether or not an individual may develop PD include environment and genetic (biologic, hereditary) factors. Studies have show that certain things may be triggers, for example cells in the brain that are made active and associated inflammation in the brain. The gut is the largest interface between the PD patient and the environment, and it is highly thought to be pathway to the environment trigger. Research studies have looked at how information is passed back and forth between the brain and the gut.

The goal of this study (pilot) is to gather information to conduct a larger clinical trial. For this pilot study is to determine if a microbiota-directed (bacteria in the gut) intervention (dietary bar) is capable of correcting the bacteria gut balance in PD. This is based on the thought that an imbalance of bacteria in the gut of PD patients may lead to the gut and intestines working correctly. The long term goal is to see if the intervention has the potential to modify the disease or protect the brain in PD. If the intervention successfully improves the bacterial imbalance in PD, it will be the first attempt to modify the Gut-Brain communication in PD, which can lead to additional studies aimed at improving the disease progression or prevention.

In this project, the investigators will test how well Parkinson's disease patients tolerate changes in the gut and intestines by providing the participants a dietary bar to eat for 10 days. The investigators intend to conduct this pilot clinical trial in which the investigators believe that daily oral intake of a "prebiotic" mixture will be safe and well tolerated in a small number Parkinson's disease participants prior to a larger clinical trial looking at efficacy.

DETAILED DESCRIPTION:
Intestinal microbiota, are a dynamic community of commensal bacteria that modulate gut homeostasis and systemic biological processes including brain development and function through a bidirectional "Gut-Brain axis". Recent studies in both rodent models of disease and human have shown disrupted intestinal microbiota community in multiple systemic metabolic and inflammatory disorders including neurological disease. More specifically emerging evidence shows that stool and intestinal mucosal associated microbiota composition and function are abnormal in PD patients. Divergence of commensal bacteria composition from the microbial communities found in healthy persons (so called "dysbiosis"), has been associated with PD in early and late stages, as well as in patients with Rapid Eye Movement (REM) sleep behavior disorder (RBD), a group that are at high risk of progression to PD.

In this project, the investigators will test the tolerability of Parkinson's disease patients in modulating the gut microbiota through dietary means. The investigators intend to conduct a pilot clinical trial in which the investigators hypothesize that daily oral intake of a prebiotic mixture will be safe and well tolerated in a small number Parkinson's disease participants prior to a larger clinical trial looking at efficacy.

Research design and protocol:

The study is an open-label, non-randomized study in 20 Parkinson's disease participants at Rush University Medical Center (RUMC) under the supervision of Drs. Hall and Keshavarzian. The trial will include 10 PD patients who are de novo (not yet on medication) or moderate stage (on medications). Participants will take the prebiotics in a form of a bar (Table 1) for 10 days- one bar (10 gram fiber) a day for 3 days and then one bar twice a day for additional one week.

Each participant will have a baseline visit and a follow up visit after 10 days of the intervention (consumption of prebiotic dietary bar). At each visit, participants will complete questionnaires regarding adverse events including a questionnaire that rates bowel movement, stool consistency, discomfort, flatulence, abdominal pain, and bloating on a scale from 1 (best) to 10 (worst). Participants will also complete a Perceived Stress Questionnaire (Appendix D) and GI Symptom and Severity Checklist (Appendix A). Participants will be asked to fill out a diet record (24ASA diet questionnaire) (Appendix E) during the last 3 days on the intervention. Participant will also are asked to self-collect stool at home before consuming (eating) the first probiotic bar in the study and during the last day of the study at home. Supplies for stool collection (2 stool collection kit) and instructions for specimen handling and for completing these tasks will be given at Visit 1 and refreshed before visit 2. At visit 1 participants will be provided with 2 stool collection kits. First stool will be collected at home about 1 day and participants are asked to mail the stool in a pre-paid Fed Ex right after collecting the stool. The second stool collection will be on the last day that participants consume the probiotic bars prior to coming to for study visit 2 when the participants bring the stool to the study visit. The kit includes supplies to preserve the sample with gas packs and collection bag so the sample can be brought with the participant to the visits within 24 hours. The self-collected stool samples will be saved by the study team and frozen for future use. Participants will be asked to complete several dietary questionnaires including a Mediterranean diet screener (Appendix F), food timing screener (Appendix B) and food frequency questionnaire (Appendix C). Before Visit 2, each participant will collect the stool and complete the 3-day food record; these will be returned at Visit 2. At Visit 2, participants will complete a Perceived Stress Questionnaire (Appendix D) and GI Symptom and Severity Checklist and associated instructions (Appendix A). Each participant will also have blood draw (1 red top to collect serum and 1 EDTA tube to collect plasma) at visit 1 (baseline) and at visit 2 (completion of the study) to check for serum short chain fatty acids, lipopolysaccharides, interleukins and cytosine monophosphate(check for safety).

Participants will provide written informed consent (Visit 1) before any study procedures, data or sample collection are performed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease,
* >age 30,
* Must be able to consent

Exclusion Criteria:

* prior intestinal resection,
* patient history of GI diseases except for hiatal hernia, gastroesophageal reflux disease, hemorrhoids,
* severe renal disease defined by creatinine more than 2 ½ times normal,
* markedly abnormal liver function defined by liver function tests over 4 times normal levels or elevated bilirubin,
* antibiotic use within the last 12 weeks prior to enrollment,
* a plan to have a major change in dietary habit during the study,
* consumption of probiotics, prebiotics or synbiotics without an appropriate 2 week washout period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Tolerability of prebiotic bar after 10 days in PD participants | 10 days
  Tolerability of the prebiotic bar will be assessed for change in the GI Symptoms and Severity Checklist at 10 days from baseline

SECONDARY OUTCOMES:
Safety of prebiotic bar during 10 days in Parkinson's disease participants | 10 days
  Measurement of safety will be assessed using the frequency of adverse events over the 10 day trial period

OTHER OUTCOMES:
Changes in the relative abundance of SCFA-producing bacteria | 10 days
  SCFA analysis will be performed on the blood collected
Changes in intestinal barrier integrity | 10 days
  Zonulin and LBP/LPS
Changes in brain health | 10 days
  neurofilament light chain
Changes in PD related gastrointestinal symptoms | 10 days
  GI Questionnaires
Changes in intestinal systemic inflammation | 10 days
  Serum Cytokines and stool calprotectin

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Hall, MD PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Cener, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall DA, Voigt RM, Cantu-Jungles TM, Hamaker B, Engen PA, Shaikh M, Raeisi S, Green SJ, Naqib A, Forsyth CB, Chen T, Manfready R, Ouyang B, Rasmussen HE, Sedghi S, Goetz CG, Keshavarzian A. An open label, non-randomized study assessing a prebiotic fiber intervention in a small cohort of Parkinson's disease participants. Nat Commun. 2023 Feb 18;14(1):926. doi: 10.1038/s41467-023-36497-x. PMID 36801916